CLINICAL TRIAL: NCT01427231
Title: The Short-term Effect of Glucose and Sacharose Ingestion on Cognitive Performance and Mood in Elderly Subjects
Brief Title: Short-term Effect of Glucose and Sacharose Ingestion on Cognitive Performance and Mood in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Suikerstichting Nederland (Baarn) (Unknown)
Responsible Party: Principal Investigator, Lisette de Groot, PhD, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: NL36813.081.11
Record Dates: First submitted 2011-08-26; First posted 2011-09-01 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Mental Health; Cognition; Memory; Attention
Keywords: Cognitive performance; Attention; Memory; Glucose; Sacharose; Elderly; Memory complaints
MeSH Terms: conditions — Psychological Well-Being | interventions — Glucose; Sucrose; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Drink with 50 g glucose (Active Comparator): The glucose drink contains 50 g of glucose soluted in 250 ml of water and lemon juice.
  Interventions: Dietary Supplement: glucose
- Drink with 100 gram of sacharose (Active Comparator): The sacharose drink contains 100 g of sacharose soluted in 250 ml of water and lemon juice.
  Interventions: Dietary Supplement: sacharose
- Placebo with sweeteners (Placebo Comparator): The placebo contains a mixture of artificial sweeteners in order to have the same sweetness and appearance of the test drinks (the glucose drink and the sacharose drink).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: glucose — The effect of a glucose solution on cognitive performance will be measured.
  Other Names: Sucrose, sugar.
  Arms: Drink with 50 g glucose
Dietary Supplement: sacharose — The effect of a sacharose solution on cognitive performance will be measured.
  Arms: Drink with 100 gram of sacharose
Dietary Supplement: Placebo — The effect of a placebo drink with sweeteners on cognitive performance will be measured.
  Arms: Placebo with sweeteners

SUMMARY:
The objective of the current study is to determine the acute effect of a glucose drink and a sacharose drink compared to a placebo on cognitive performance in elderly with light memory complaints. The investigators expect that the sugar containing drinks will improve memory and attentional functions. Furthermore, blood glucose response will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 70 years and older
* Memory complaints

Exclusion Criteria:

* Type I or II diabetes
* Parkinson disease
* MMSE < 25 (to exclude cognitively impaired subjects
* CES-D > 16 (to exclude depressive subjects)
* Pharmacological antidepressives or medication for dementia
* Liver disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Performance on the paired associate recall test | cognitive tests will start 15 minutes after ingestion of the intervention product
  Cognitive performance will be assessed by several sensitive tests. Power is calculated on the paired associate recall test, but also several other cognitive performance test focusing on memory, attention and reaction time will be performed

SECONDARY OUTCOMES:
Mood | within 15 minutes after consuming the test drink and after completing the cognitive tests (within 90 minutes after consuming the test drink)
  Mood will be measured by the POMS, after consuming the test drink, and after completing the congitive tests.
Blood glucose response | from baseline till 90 minutes after consuming the drink
  Blood glucose will be measured at five time points, at t=0, after 15 minutes, 30, 60 and 90 minutes.
Plasma insulin levels | At t= -15 minutes, before consuming the test drink
  One venapunction will be carried out at baseline to measure plasma insulin levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands